CLINICAL TRIAL: NCT02959567
Title: Effectiveness and Safety Evaluation of Aqueduct 100-device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aqueduct Medical Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AQD 01-04
Record Dates: First submitted 2016-11-02; First posted 2016-11-09 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: Cervix Uteri Dilation
Keywords: cervix; cervical dilation; balloon catheter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aqueduct 100 dilation (Experimental): Uterine cervix dilation through Aqueduct-100 device
  Interventions: Device: Aqueduct 100 dilation

INTERVENTIONS:
Device: Aqueduct 100 dilation

SUMMARY:
Evaluation of efficacy and safety of using Aqueduct -100 - Cervical Dilator Device, focusing on diagnostic or operative hysteroscopies.

DETAILED DESCRIPTION:
There are predominantly two major dilatation techniques that are employed in dilating the cervix. The first technique uses expansible dry solid material, such as laminaria (seaweed) is inserted into the cervix in its dried stiff form. In the cervix it comes into contact with body fluids that cause the laminaria to swell and enlarge the cervical cavity. The second more widespread procedure, involves the use of series of solid, rod like instruments of graduated diameter used in serial fashion by the physician (Hegar dilators). The physician first inserts a rod like dilator and replaces it with the dilator of next higher diameter. This procedure continues until adequate dilatation occurs.

The Problem is that each of the above-mentioned methods has its shortcomings: the use of the laminaria method (rarely done) requires preliminary patient visit, for insertion of the laminaria rod and is extremely slow and typically involves often as much as 10-12 hours for a significant amount of dilatation to occur.

The use of rod-like instruments (Hegar) requires general or regional anesthesia, when local anesthetics are used, the patient nevertheless frequently experiences a great amount of discomfort from the procedure. The mechanical dilatation of the cervix demands a large amount of longitudinal force that may damage or even puncture the cervix and the uterus.

Aqueduct 100 is a catheter for use in dilating various body cavities and especially the human cervix. The device will enable continuous, fast and safe dilatation of the cervix to a pre-determined diameter as a pre-procedure to intrauterine surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Subjects, females, 18 years of age or older.
* Subjects undergoing diagnostic or operative hysteroscopies
* Subjects willing to sign informed consent form.

Exclusion Criteria:

* Subjects younger than 18 years of age
* Subjects unwilling to sign the informed consent form
* Pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients in which, through 1 minute dilation with Aqueduct-100, a cervix dilation of 5mm, required for diagnostic/ operative hysteroscopy, is reached. | Through study completion, an average of 11 months
  Efficacy evaluation of Aqueduct-100
Occurrence of Adverse Events | Through study completion, an average of 11 months
  In vivo safety evaluation of using Aqueduct-100

SECONDARY OUTCOMES:
Measurement of physicians'overall satisfaction with the device, through a questionnaire | Through study completion, an average of 11 months

CONTACTS AND LOCATIONS:
Overall Officials: Larry Spiegelman, Dr., Principal Investigator — Baptist Medical Arts Surgical Center
Locations (1):
- Baptist Medical Arts Surgical Center, Gynecology Department, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mazza E, Nava A, Bauer M, Winter R, Bajka M, Holzapfel GA. Mechanical properties of the human uterine cervix: an in vivo study. Med Image Anal. 2006 Apr;10(2):125-36. doi: 10.1016/j.media.2005.06.001. Epub 2005 Sep 6. PMID 16143559
- [Background] Buhimschi, C.; Buhimschi, I.; Malinow, A.; Saade, G.; Garfield, R.; Weiner, C., The Forces of Labour. Fetal and Maternal Medicine Review 2003, 14 (4), 273-307.
- [Background] Myers KM, Paskaleva AP, House M, Socrate S. Mechanical and biochemical properties of human cervical tissue. Acta Biomater. 2008 Jan;4(1):104-16. doi: 10.1016/j.actbio.2007.04.009. Epub 2007 Sep 27. PMID 17904431
- [Background] Kenyon NJ, Stevens JC, Stewart P, Black MM, Clifford A. A critical investigation of the measurement of the force required to dilate the human uterine cervix. Clin Phys Physiol Meas. 1988 May;9(2):155-61. doi: 10.1088/0143-0815/9/2/008. PMID 3391017
- [Background] S. Febvay, S. Socrate and M.D. House. Biomechanical modeling of cervical tissue. A quantitative investigation of cervical funneling. Proceedings of the ASME 2003 International Mechanical Engineering Congress and Exposition, Washington, D.C., November 2003.
- [Background] Arsenijevic S, Vukcevic-Globarevic G, Volarevic V, Macuzic I, Todorovic P, Tanaskovic I, Mijailovic M, Raicevic S, Jeremic B. Continuous controllable balloon dilation: a novel approach for cervix dilation. Trials. 2012 Oct 22;13:196. doi: 10.1186/1745-6215-13-196. PMID 23088906
- [Background] Nicolaides KH, Welch CC, MacPherson MB, Johnson IR, Filshie GM. Lamicel: a new technique for cervical dilatation before first trimester abortion. Br J Obstet Gynaecol. 1983 May;90(5):475-9. doi: 10.1111/j.1471-0528.1983.tb08947.x. PMID 6849849